CLINICAL TRIAL: NCT05326295
Title: Surveillance of Circulating Tumor Cell Phenotype in Early Stage Breast Cancer Patients With Neoadjuvant Chemotherapy or Adjuvant Chemotherapy
Brief Title: Evaluation of Treatment Efficacy by Circulating Tumor Cell Phenotype Surveillance in Breast Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: Hunan Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KYJJ-2021-186
Record Dates: First submitted 2022-03-16; First posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-03

CONDITIONS: Breast Neoplasms; Neoplastic Cells, Circulating; Chemotherapy Effect
MeSH Terms: conditions — Breast Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Breast cancer patients
  Interventions: Diagnostic Test: CTC detection

INTERVENTIONS:
Diagnostic Test: CTC detection — CTCs separation and enrichment technology. Combined with the prognosis of patients with recurrence and survival time, we explored the evaluation of CTC number, cell phenotype distribution, PDL1 and FOXC2 expression on the prognosis of early stage breast cancer patients. The research results are expected to provide a new effective index and theoretical basis for evaluating the treatment efficacy of breast cancer patients.

SUMMARY:
The phenotype of circulating tumor cells (CTCs) is supposed to be significant indicator that is correlated the prognosis of breast cancer patients who have completed neoadjuvant chemotherapy, primary tumor surgery with/without adjuvant chemotherapy. The aim of this observational study is to assess the efficacy of CTCs surveillance in predicting the prognosis of breast cancer patients.

DETAILED DESCRIPTION:
The aim of this observational study is to assess the efficacy of CTCs surveillance in predicting the treatment response of neoadjuvant chemotherapy, surgery and adjuvant chemotherapy. This study also aims to evaluate the efficacy of CTCs surveillance in predicting invasive-disease free survival (iDFS), overall survival (OS) and metastasis. Additionally, this study evaluate the expression of PDL1 and FOXC3 on CTCs.

ELIGIBILITY:
Inclusion Criteria

* The age is more than 18 years old;
* Pathology confirmed malignant breast tumor;
* No clinical diagnosis of other malignancies, unstable complications or uncontrolled infection;
* Life expectancy is greater than 6 month;
* The main organ function is normal;
* The subjects volunteered to participate in this study, signed informed consent, followed up with good compliance.

Exclusion Criteria

* Patients who had suffered from other malignant tumors;
* With uncontrolled bacterial, viral or fungal infections;
* With physical or mental disorders
* Without or limited civil capacity;
* Infected with human immunodeficiency virus (HIV)；
* Circumstances in which the investigator considers it inappropriate to participate in this study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Early stage breast cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
iDFS | From date of enrollment through study completion, up to 10 years.
  The survival time from the date of tumor resection to the date of the relapse of the invasive disease.

SECONDARY OUTCOMES:
overall survival | From date of enrollment through study completion, up to 10 years.
  The survival time from the date of recruitment to the date of death.
Pathological complete response rate | From date of enrollment up to 24 weeks
  pCR is defined as no infiltrating tumor cells in pathological examination in the primary breast and axillary lymph nodes.

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China